CLINICAL TRIAL: NCT02017730
Title: An Open-Label Study To Evaluate The Safety and Tolerability Of A Novel LPA1 Receptor Positron Emission Tomography (PET) Ligand [11C]BMT-136088 And To Assess Receptor Occupancy In Human Lung Following Oral Administration Of BMS-986020 In Healthy Subjects
Brief Title: To Evaluate The Relationship Between Plasma Drug Levels And Receptor Binding in Lung Using PET (Positron Emission Tomography) In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IM136-106
Record Dates: First submitted 2013-12-17; First posted 2013-12-23 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Immunology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Part 1: [11C]BMT-136088 (Safety Study) (Experimental): Single PET SCAN with single bolus injection of [11C]BMT-136088
  Interventions: Drug: [11C]BMT-136088
- Part 2: [11C]BMT-136088 (Test/Retest study) (Experimental): Single PET SCAN with Intravenous (IV) bolus plus infusion of [11C]BMT-136088 followed by a re-test PET scan (approximately 6 hours apart) with IV bolus plus infusion of [11C]BMT-136088
  Interventions: Drug: [11C]BMT-136088
- Part 3: BMS-986020+[11C]BMT-136088 (Receptor Occupancy study) (Experimental): BMS-986020 Tablets or Oral Solution of 4 dose levels from from the 6 dose levels of (50 mg, 150 mg, 300 mg, 600 mg, 1200 mg and 1500 mg) and 3 PET SCANS (Pre-Dose, Post-Dose1, Post-Dose2) with bolus plus infusion of [11C]BMT-136088
  Interventions: Drug: BMS-986020; Drug: [11C]BMT-136088
- Part 4: [11C]BMT-136088 (Tissue Distribution study) (Experimental): Single PET SCAN with [11C]BMT-136088 to evaluate additional tracer uptake sites in humans other than the lung, such as heart, kidney, liver, gallbladder, etc.
  Interventions: Drug: [11C]BMT-136088

INTERVENTIONS:
Drug: BMS-986020
  Arms: Part 3: BMS-986020+[11C]BMT-136088 (Receptor Occupancy study)
Drug: [11C]BMT-136088

SUMMARY:
The purpose of this study is to assess the safety and tolerability of a novel positron emission tomography (PET) tracer [11C]BMT-136088 in healthy adult subjects for measurement of availability of Lysophosphatidic Acid (LPA1) receptors in the human lung and to use this tracer to assess LPA1 receptor occupancy using [11C]BMT-136088 in the human lung following oral administration of Bristol Myers Squibb (BMS)-986020.

DETAILED DESCRIPTION:
End point Classification: Pharmacokinetics/Pharmacodynamics

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Body weight at least 50kg (110lbs), Body Mass Index (BMI) within 19 to 32 kg/m2, inclusive
* Must be in good health as determined by medical history, physical examination, ECG, serum/urine biochemistry, hematology, and serology tests
* Negative hepatitis panel and negative human immunodeficiency virus (HIV)antibody screens

Exclusion Criteria:

* Any history or presence of clinically significant respiratory, Gastro Intestinal (GI), renal, hepatic, pancreatic, hematological, neurological (including history of seizure), cardiovascular, psychiatric (including known addictive disorders), musculoskeletal, genitourinary, immunological, or dermatological disorders, including all cancers
* Any acute or chronic condition that, in the opinion of the investigator in consultation with the BMS Medical Monitor, could jeopardize the subject's safety, tolerability, or pharmacokinetics of the BMS-986020
* Any major surgery within 4 weeks of study drug administration
* Existence of a cold, upper respiratory tract infection, or fever within 5 days prior to check-in
* Presence or history of any abnormality or illness that may affect absorption, distribution, metabolism or elimination of the study drug
* Donation of blood or plasma (exclude the screening visit) within 2 months prior to check in through end of synthesis (EOS), inclusive

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Overall safety and tolerability of novel tracer [11C]BMT-136088 | Approximately up to 90 days
  The following safety endpoints will be considered, the incidence of adverse events (AEs), serious AEs, AEs leading to discontinuation from the study, and death as well as marked abnormalities in clinical laboratory tests, vital sign measurements, electrocardiograms (ECGs), and physical examinations occurring from screening up to study discharge.
Lung LPA1 percentage receptor occupancy of BMS-986020 | Up to 2 days post BMS-986020 administration
  Assessed by [11C]BMT-136088 tracer lung volume of distribution (VT) before and after single oral dose of BMS-986020.

SECONDARY OUTCOMES:
Exposure-response relationship between lung LPA1 percentage receptor occupancy and BMS-986020 plasma concentration. | Up to 48 hr postdose (Approximately up to Day 3)
Maximum observed concentration (Cmax) of BMS-986020 | 13 timepoints up to Day 3
Time of maximum observed concentration (Tmax) of BMS-986020 | 13 timepoints up to Day 3
Area under the concentration-time curve from time zero to the time of the last quantifiable concentration [AUC(0-T)] of BMS-986020 | 13 timepoints up to Day 3
Area under the concentration-time curve from time zero extrapolated to infinite time [AUC(INF)] of BMS-986020 | 13 timepoints up to Day 3
Half life (T-HALF) of BMS-986020 | 13 timepoints up to Day 3
Safety of single oral dose of BMS-986020 where [11C]BMT-136088 is administered to healthy subjects | Approximately up to 90 days
  Safety based on incidence of AEs, serious AEs, AEs leading to discontinuation, and death as well as marked abnormalities in clinical laboratory tests, vital sign measurements, ECGs, and physical examinations

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Yale Pet Center, New Haven, Connecticut, United States

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx